CLINICAL TRIAL: NCT04433936
Title: Corneal Tomographic Analysis Among Patients With Thyroid Gland Dysfunction.
Brief Title: Corneal Tomographic Parameters in TGD
Status: Completed | Type: Observational
Sponsor: Ameera Gamal Abdelhameed (Other)
Responsible Party: Sponsor-Investigator, Ameera Gamal Abdelhameed, Lecturer of Ophthalmology, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: Pentacam parameters in TGD
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Keratoconus; Corneal Ectasia; Thyroid Eye Disease
Keywords: keratoconus; pentacam; TED
MeSH Terms: conditions — Keratoconus; Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid Gland Dysfunction: Patients with a recent diagnosis of TGD (the study group) were recruited from endocrinology outpatient clinic of Specialized Medical Hospital, Mansoura University. Diagnosis of TGD was based on précised history, clinical examination and laboratory investigations. In order to avoid bias, patients with history of intake of any thyroid-related medications (antithyroid medications or thyroxine replacement), radioactive iodine or thyroidectomy were excluded from the study.
  Interventions: Diagnostic Test: Pentacam tomography
- Control: fifty age and gender matched healthy subjects without known personal or family history of thyroid disease or any autoimmune diseases were recruited from candidates of refractive surgery referred to the outpatient clinic of Mansoura Ophthalmology Center for pentacam assessment and who were proved to have normal corneal pentacam parameters. They were further examined by the endocrinologist to exclude thyroid dysfunction; this was supported by normal thyroid function profile (serum TSH and free T4) and negative anti-TPO and antithyroglobulin antibodies.
  Interventions: Diagnostic Test: Pentacam tomography

INTERVENTIONS:
Diagnostic Test: Pentacam tomography — The Pentacam maps were analyzed. The following anterior and posterior corneal surface parameters were evaluated by the Scheimpflug system: Kf, Ks, Kmax. The pachymetric map was analyzed, including CCT at the apex of the geometric center and CTmin. PPIavg, PPI min and PPI max were calculated . The Ambrósio relational thickness (ART) was calculated The posterior corneal elevation maps were evaluated and the posterior corneal elevation values relative to this reference were recorded. The back difference elevation and multimetric D index values were extrapolated from the difference map of the Belin/Ambrósio-enhanced ectasia display of the Pentacam system.

SUMMARY:
The current study involved analysis of the corneal tomographic parameters of patients with thyroid gland dysfunction (hyperthyroidism or hypothyroidism), including those with an autoimmune etiology, in comparison to healthy controls without TGD, using pentacam, in an attempt to detect possible early corneal changes and to highlight whether early screening of those patients would be necessary for early detection of KC.

DETAILED DESCRIPTION:
A total of 100 eyes of 50 patients with TGD and 100 eyes of 50 healthy controls were enrolled. Diagnosis of TGD was based on history, clinical examination and laboratory investigations. Exclusion criteria included previous thyroid medications, thyroidectomy, previous ocular surgery, corneal pathology and other risk factors of keratoconus (KC). All eyes were examined by Pentacam, (Oculus Optikgerate GmbH, Wetzlar, Germany). Pentacam parameters were compared between TGD patients and controls. Spearman's correlation coefficient between different pentacam parameters and the level of free T4 and TSH was calculated.

ELIGIBILITY:
Inclusion Criteria:

* For TGD patients: Patients with a recent diagnosis of TGD (the study group) were recruited from endocrinology outpatient clinic of Specialized Medical Hospital, Mansoura University. Diagnosis of TGD was based on précised history, clinical examination and laboratory investigations. In order to avoid bias, patients with history of intake of any thyroid-related medications (antithyroid medications or thyroxine replacement), radioactive iodine or thyroidectomy were excluded from the study. Therefore, we only included patients who did not received treatment yet For the control group, fifty age and gender matched healthy subjects without known personal or family history of thyroid disease or any autoimmune diseases were recruited from candidates of refractive surgery referred to the outpatient clinic of Mansoura Ophthalmology Center for pentacam assessment and who were proved to have normal corneal pentacam parameters. They were further examined by the endocrinologist to exclude thyroid dysfunction; this was supported by normal thyroid function profile (serum TSH and free T4) and negative anti-TPO and antithyroglobulin antibodies.

Exclusion Criteria:

* patients with previous thyroid medications or replacement therapy, thyroidectomy or radioactive iodine intake participants with a history of ocular surgery or trauma, use of any topical medication or contact lens wear, patients with any corneal pathology, Corneal dystrophy, corneal scarring or any concurrent ocular disease. To eliminate other risk factors for KC, we also excluded participants with a history of persistent eye rubbing, vernal keratoconjunctivitis (VKC), atopy, Down syndrome, Turner's syndrome, or congenital rubella. Pregnant or lactating females were also excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 eyes of 50 patients with TGD (hypo-hyperthyroidism) and 100 eyes of 50 age and sex matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
corneal tomographic parameter | 1 day (once at first recruitment)
  analysis of pentacam maps

CONTACTS AND LOCATIONS:
Overall Officials: Rania Bassiouny, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Davidson AE, Hayes S, Hardcastle AJ, Tuft SJ. The pathogenesis of keratoconus. Eye (Lond). 2014 Feb;28(2):189-95. doi: 10.1038/eye.2013.278. Epub 2013 Dec 20. PMID 24357835
- [Background] McMonnies CW. Inflammation and keratoconus. Optom Vis Sci. 2015 Feb;92(2):e35-41. doi: 10.1097/OPX.0000000000000455. PMID 25397925
- [Background] Galvis V, Sherwin T, Tello A, Merayo J, Barrera R, Acera A. Keratoconus: an inflammatory disorder? Eye (Lond). 2015 Jul;29(7):843-59. doi: 10.1038/eye.2015.63. Epub 2015 May 1. PMID 25931166
- [Background] Conrad AH, Zhang Y, Walker AR, Olberding LA, Hanzlick A, Zimmer AJ, Morffi R, Conrad GW. Thyroxine affects expression of KSPG-related genes, the carbonic anhydrase II gene, and KS sulfation in the embryonic chicken cornea. Invest Ophthalmol Vis Sci. 2006 Jan;47(1):120-32. doi: 10.1167/iovs.05-0806. PMID 16384953
- [Background] COULOMBRE AJ, COULOMBRE JL. CORNEAL DEVELOPMENT. 3. THE ROLE OF THE THYROID IN DEHYDRATION AND THE DEVELOPMENT OF TRANSPARENCY. Exp Eye Res. 1964 Jun;3:105-14. doi: 10.1016/s0014-4835(64)80024-5. No abstract available. PMID 14211912
- [Background] Robson H, Siebler T, Stevens DA, Shalet SM, Williams GR. Thyroid hormone acts directly on growth plate chondrocytes to promote hypertrophic differentiation and inhibit clonal expansion and cell proliferation. Endocrinology. 2000 Oct;141(10):3887-97. doi: 10.1210/endo.141.10.7733. PMID 11014246
- [Background] Kocak Altintas AG, Gul U, Duman S. Bilateral keratoconus associated with Hashimoto's disease, alopecia areata and atopic keratoconjunctivitis. Eur J Ophthalmol. 1999 Apr-Jun;9(2):130-3. doi: 10.1177/112067219900900210. PMID 10435426
- [Background] Thanos S, Oellers P, Meyer Zu Horste M, Prokosch V, Schlatt S, Seitz B, Gatzioufas Z. Role of Thyroxine in the Development of Keratoconus. Cornea. 2016 Oct;35(10):1338-46. doi: 10.1097/ICO.0000000000000988. PMID 27560028
- [Background] Flasko Z, Zemova E, Eppig T, Modis L, Langenbucher A, Wagenpfeil S, Seitz B, Szentmary N. Hypothyroidism is Not Associated with Keratoconus Disease: Analysis of 626 Subjects. J Ophthalmol. 2019 Oct 31;2019:3268595. doi: 10.1155/2019/3268595. eCollection 2019. PMID 31815013
- [Background] El-Massry A, Doheim MF, Iqbal M, Fawzy O, Said OM, Yousif MO, Badawi AE, Tawfik A, Abousamra A. Association Between Keratoconus and Thyroid Gland Dysfunction: A Cross-Sectional Case-Control Study. J Refract Surg. 2020 Apr 1;36(4):253-257. doi: 10.3928/1081597X-20200226-03. PMID 32267956
- [Background] Alhawari HH, Khader YS, Alhawari HH, Alomari AF, Abbasi HN, El-Faouri MS, Al Bdour MD. Autoimmune Thyroid Disease and Keratoconus: Is There an Association? Int J Endocrinol. 2018 Jul 31;2018:7907512. doi: 10.1155/2018/7907512. eCollection 2018. PMID 30154844
- [Background] Karabulut GO, Kaynak P, Altan C, Ozturker C, Aksoy EF, Demirok A, Yilmaz OF. Corneal biomechanical properties in thyroid eye disease. Kaohsiung J Med Sci. 2014 Jun;30(6):299-304. doi: 10.1016/j.kjms.2014.02.015. Epub 2014 Apr 17. PMID 24835350
- [Background] Moghimi S, Safizadeh M, Mazloumi M, Hosseini H, Vahedian Z, Rajabi MT. Evaluation of Corneal Biomechanical Properties in Patients With Thyroid Eye Disease Using Ocular Response Analyzer. J Glaucoma. 2016 Mar;25(3):269-73. doi: 10.1097/IJG.0000000000000254. PMID 26020688
- [Background] Kirgiz A, Cabuk KS, Yetmis M, Atalay K. Corneal biomechanical properties in patients with Hashimoto's thyroiditis. Adv Clin Exp Med. 2019 Jan;28(1):109-112. doi: 10.17219/acem/85039. PMID 30311752
- [Background] Gatzioufas Z, Panos GD, Brugnolli E, Hafezi F. Corneal topographical and biomechanical variations associated with hypothyroidism. J Refract Surg. 2014 Feb;30(2):78-9. doi: 10.3928/1081597X-20140120-01. No abstract available. PMID 24477035
- [Background] UTIGER RD. RADIOIMMUNOASSAY OF HUMAN PLASMA THYROTROPIN. J Clin Invest. 1965 Aug;44(8):1277-86. doi: 10.1172/JCI105234. No abstract available. PMID 14322035
- [Background] Ross DS, Burch HB, Cooper DS, Greenlee MC, Laurberg P, Maia AL, Rivkees SA, Samuels M, Sosa JA, Stan MN, Walter MA. 2016 American Thyroid Association Guidelines for Diagnosis and Management of Hyperthyroidism and Other Causes of Thyrotoxicosis. Thyroid. 2016 Oct;26(10):1343-1421. doi: 10.1089/thy.2016.0229. PMID 27521067
- [Background] Chaudhary V, Bano S. Thyroid ultrasound. Indian J Endocrinol Metab. 2013 Mar;17(2):219-27. doi: 10.4103/2230-8210.109667. PMID 23776892
- [Background] Ambrosio R Jr, Caiado AL, Guerra FP, Louzada R, Sinha RA, Luz A, Dupps WJ, Belin MW. Novel pachymetric parameters based on corneal tomography for diagnosing keratoconus. J Refract Surg. 2011 Oct;27(10):753-8. doi: 10.3928/1081597X-20110721-01. Epub 2011 Jul 29. PMID 21800785
- [Background] O'Brart DP, Patel P, Lascaratos G, Wagh VK, Tam C, Lee J, O'Brart NA. Corneal Cross-linking to Halt the Progression of Keratoconus and Corneal Ectasia: Seven-Year Follow-up. Am J Ophthalmol. 2015 Dec;160(6):1154-63. doi: 10.1016/j.ajo.2015.08.023. Epub 2015 Aug 22. PMID 26307513
- [Background] Bahceci UA, Ozdek S, Pehlivanli Z, Yetkin I, Onol M. Changes in intraocular pressure and corneal and retinal nerve fiber layer thicknesses in hypothyroidism. Eur J Ophthalmol. 2005 Sep - Oct 2005;15(5):556-561. doi: 10.5301/EJO.2008.1004. PMID 28221458
- [Background] Gatzioufas Z, Thanos S. Acute keratoconus induced by hypothyroxinemia during pregnancy. J Endocrinol Invest. 2008 Mar;31(3):262-6. doi: 10.1007/BF03345600. PMID 18401210
- [Background] Hoogewoud F, Gatzioufas Z, Hafezi F. Transitory topographical variations in keratoconus during pregnancy. J Refract Surg. 2013 Feb;29(2):144-6. doi: 10.3928/1081597X-20130117-11. PMID 23380417
- [Background] Hafezi F, Iseli HP. Pregnancy-related exacerbation of iatrogenic keratectasia despite corneal collagen crosslinking. J Cataract Refract Surg. 2008 Jul;34(7):1219-21. doi: 10.1016/j.jcrs.2008.02.036. PMID 18571094
- [Background] Lang GE, Naumann GO. [Keratoconus in Alagille syndrome]. Klin Monbl Augenheilkd. 1991 Jun;198(6):555-7. doi: 10.1055/s-2008-1046031. German. PMID 1895727
- [Background] 27. King EF. Keratoconus following thyroidectomy. Transactions of the Ophthalmological Societies of the United Kingdom. 1953; 73: 31-39.
- [Background] Lee R, Hafezi F, Randleman JB. Bilateral Keratoconus Induced by Secondary Hypothyroidism After Radioactive Iodine Therapy. J Refract Surg. 2018 May 1;34(5):351-353. doi: 10.3928/1081597X-20171031-02. PMID 29738593
- [Background] Ucakhan OO, Cetinkor V, Ozkan M, Kanpolat A. Evaluation of Scheimpflug imaging parameters in subclinical keratoconus, keratoconus, and normal eyes. J Cataract Refract Surg. 2011 Jun;37(6):1116-24. doi: 10.1016/j.jcrs.2010.12.049. PMID 21596255
- [Background] 30. Baker KC, Chen YL, Shi L, Lewis JWL, Kugler L, Wang M. Does the Posterior Corneal Elevation Provide the First Indication of Keratoconus? Invest. Ophthalmol. Vis. Sci. 2010; 51(13):4963.
- [Background] Nemet AY, Vinker S, Bahar I, Kaiserman I. The association of keratoconus with immune disorders. Cornea. 2010 Nov;29(11):1261-4. doi: 10.1097/ICO.0b013e3181cb410b. PMID 20802320
- [Background] AlHawari HH and Al Bdour MD. Vernal keratoconjunctivitis and severe keratoconus associated with autoimmune polyglandular syndrome type II (APS-2): a case report," Jordan Medical Journal 2016; 50(3): 157-159.